CLINICAL TRIAL: NCT06847581
Title: JAME: Hand Tremor Recognition and Control Based on Accelerometers and Non-invasive Electrical Stimulation. A Pilot Feasibility Study on PD and ET Patients.
Brief Title: JAME, a Wearable Device to Control Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JAME2020
Record Dates: First submitted 2024-03-07; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease; Essential Tremor
Keywords: parkinson's disease, essential tremor, transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Intervention Model Description: open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parkinson'Disease (Experimental): Patients with Parkinson's disease with resting tremor alone at the start of their disease
  Interventions: Device: JAME
- Essential Tremor (Experimental): Patients with Essential Tremor
  Interventions: Device: JAME

INTERVENTIONS:
Device: JAME — JAME is a wearable device able to monitor movements of the upper limbs and, through an ad-hoc algorithm based on machine learning, can recognize tremor and suppress it through TENS

SUMMARY:
The study is a pilot feasibility study aimed at verifying that (1) tremor can be recognized using an accelerometer placed on the hand area and a data mining algorithm properly trained and (2) TENS applied in the hand area is able to acutely suppress hand tremor respect to the baseline.

DETAILED DESCRIPTION:
The study includes 2 different groups: 9 patients with Parkinson's disease with resting tremor alone at the start of their disease (group1), and 5 patients with Essential Tremor (group2). For both groups, the study protocol includes an initial screening visit, in which, after enrollment, the patient's baseline is defined. The experimental session combines both tremor recording and a TENS stimulation treatment.

During the experimental session, the patient wears two devices able to record the upper limb's motion. These devices are commercially available wearable IMU sensors equipped with a triaxial accelerometer, a triaxial gyroscope and triaxial magnetometer. One device is located on the hand, the other on the wrist of the same upper limb, the dominant one. Patients are asked to perform the tasks of the WHIGET scale at baseline and during two different types of electrical stimulation (in a randomly assigned order).

For the recording part, the primary endpoint is the accuracy of the detection system measured as the number of correct detections of tremor episodes on the total tremor episodes recorded by the system (5 seconds windows). For the stimulation part, the primary endpoint is the reduction of upper limb tremor during the stimulation session compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed the approved Informed Consent;
* Subject is willing and able to complete the study procedures;
* Subject is ≥ 18 years of age;
* Subject has a certain diagnosis of:

  * definite PD, at the start of the disease (respecting the new International Parkinson Disease and Movement Disorder Society diagnostic criteria) and experiences tremor as measured on the UPDRS Part III; or
  * ET;
* Subject has a normal cognitive function (MMSE ≥ 24 or MoCA >26).

Exclusion Criteria:

* Atypical parkinsonian syndromes - progressive supranuclear palsy, multiple system atrophy, corticobasal degeneration, dementia with Lewy bodies, vascular Parkinsonism, and other rare causes;
* Other pre-existing and active major neurological disease;
* Pre-existing and active (e.g., on chronic medication) major psychiatric disease, such as major depression, schizophrenia, bipolar disease;
* Advanced liver, kidney, cardiac, or pulmonary disease, cancer;
* A terminal medical diagnosis consistent with survival < 1 year;
* Medical implanted devices (e.g. DBS, DUOPATM infusion pump); metal implants; the presence or even a suspicion of metal fragments or moving metal implants in its head or neck, as well as it had prior surgical operations on the head or neck;
* Dermatological lesions in the area to be treated with the electrical stimulation;
* Major drug dependency, including alcohol (in the investigator's judgment);
* Females who are pregnant or lactating;
* Subject had an important head injury in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
tremor recognition | 10 minutes
  For the recording part, the primary endpoint is the accuracy of the detection system measured as the number of correct detections of tremor episodes on the total tremor episodes recorded by the system (5 seconds windows);
tremor suppression | 10 minutes
  the primary endpoint is the reduction of upper limb tremor during the stimulation session compared to baseline, measured with the WHIGET scale

CONTACTS AND LOCATIONS:
Overall Officials: Linda Borellini, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Linda Borellini, Milan, Italy, Italy